CLINICAL TRIAL: NCT05643768
Title: Effects of Inspiratory Muscle Strength Training on Metabolic and Cardiovascular Health in Adults With Type 2 Diabetes
Brief Title: Inspiratory Muscle Strength Training in Adults With Type 2 Diabetes
Acronym: DIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 00002239
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
Keywords: insulin sensitivity; blood pressure; blood glucose; non-pharmacological; inspiratory resistance training
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated using a 1:1 ratio to A) High-Intensity Training Group (75 % maximal inspiratory pressure) or B)Low-Intensity Training Group (15% maximal inspiratory pressure)
Who Masked: Participant
Masking Description: This is a randomized trial and participants will be blinded to their allocation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-resistance IMST (Experimental): 30 breaths/day (5 sets of 6 breaths, one minute of rest between sets), 5 days/week, 6 weeks
  Interventions: Behavioral: Inspiratory muscle strength training (IMST)
- Low-resistance IMST (Active Comparator): 30 breaths/day (5 sets of 6 breaths, one minute of rest between sets), 5 days/week, 6 weeks
  Interventions: Behavioral: Inspiratory muscle strength training (IMST)

INTERVENTIONS:
Behavioral: Inspiratory muscle strength training (IMST) — 30 breaths/day, 5 days/week, 6 weeks
  Other Names: inspiratory resistance training; vascular conditioning exercise; inspiratory muscle training

SUMMARY:
This clinical research study will investigate the effects of 6 weeks of inspiratory muscle strength training on metabolic and cardiovascular outcomes in adults with recent-onset type 2 diabetes.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is at epidemic proportions in the United States and worldwide. It is a chronic obesity-associated metabolic disorder characterized by glucose dysregulation combined with insulin resistance and beta-cell defects. First-line T2DM treatments include lifestyle remedies, such as dietary modifications and exercise. Exercise, whether aerobic and/or resistance training, increases whole-body insulin sensitivity and stimulates muscle glucose uptake independent of insulin. The acute effects of exercise on muscle in patients with abnormal glucose regulation produce immediate improvements in blood glucose levels. In addition, when exercise is repeated over time, adaptations occur that include more long-lasting increases in insulin sensitivity. The effects of traditional exercise on glycemic control and insulin sensitivity in patients with T2DM are well established. However, adherence to traditional exercise programs is low, in part, due to lack of time and physical discomfort, and new regimens for T2DM treatment are needed.

Recently, a novel time-efficient respiratory exercise called Inspiratory Muscle Strength Training (IMST) was developed. IMST is distinct from other traditional forms of exercise as it is only 5 minutes per session and performed on a hand-held device during stationary sitting or standing. Typically, IMST comprises 5 sets of 6 inspiratory maneuvers with 1-minute rests between sets. Previous studies demonstrate that 6 weeks of IMST improve systolic blood pressure (SBP), sympathetic nervous system activity, and endothelial function in healthy individuals, middle-aged and older people, and adults with obstructive sleep apnea. These BP-lowering effects of IMST are significant for reducing the risks of cardiovascular disease (CVD), the number one cause of death in people living with diabetes. IMST is safe and tolerable, with adherence rates >90% in diverse populations, and presents a manageable program for improving metabolic health in T2DM patients who have difficulty maintaining a traditional exercise program requiring a large amount of time and physical exertion. It is unknown if IMST, a highly-abbreviated respiratory exercise that is not physically demanding, has beneficial effects on glycemic control and insulin sensitivity, in combination with its improvements on BP measures, in patients with T2DM. The potential for IMST to exert metabolic benefits in diabetic patients warrants assessment

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 2 diabetes by physician
* fasting plasma glucose levels ≥126 mg/dl and ≤240 mg/dl
* systolic blood pressure between 120-169 mmHg
* stable dose of medication (three months on the same dose)
* weight stable in the prior 3 months (<3.0 kg weight change) and willing to remain weight stable throughout the study
* absence of unstable clinical disease as determined by medical history

Exclusion Criteria:

* current smoker (including tobacco products, vaping devices, THC, etc…)
* have an uncontrolled medical condition (e.g., cancer)
* myocardial infarction or stroke within the previous 12 months
* performs regular aerobic exercise (>4 bouts/week)
* BMI ≥ 40 kg/m2
* systolic blood pressure <120 or ≥170 mmHg
* diastolic blood pressure >100 or <60 mmHg
* Cheyne-Stokes respiration
* history of perforated eardrum
* history of glaucoma or retinopathy
* history of collapsed lung
* diagnosed with asthma
* pregnant, breastfeeding, or trying to become pregnant (self-reported)
* medications that, in the opinion of the study physician or nurse practitioner, may impact the outcomes of the study (e.g., steroids)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline fasting blood plasma glucose after 6 weeks of IMST | Blood plasma collected and analyzed at baseline and after 6 weeks of training
  A blood sample will be collected after 12 hours of fasting. Blood and plasma will be separated and plasma glucose levels will be quantified.
Change from baseline fasting blood plasma Insulin after 6 weeks of IMST | Blood plasma collected and analyzed at baseline and after 6 weeks of training
  A blood sample will be collected after 12 hours of fasting. Blood and plasma will be separated and plasma insulin levels will be quantified.
Change from baseline insulin sensitivity after 6 weeks of IMST | Blood plasma collected and analyzed at baseline and after 6 weeks of training
  A blood sample will be collected after 12 hours of fasting. Insulin sensitivity will be calculated using the homeostatic model assessment of insulin resistance (HOMA-IR): (fasting serum insulin (mU/L) × fasting plasma glucose (mmol/L) × 22.5).

SECONDARY OUTCOMES:
Change from baseline systolic blood pressure after 6 weeks of IMST | Blood pressure will be assessed at baseline and after 6 weeks of training
  Change in systolic blood pressure (SBP) will be measured by both relative and absolute changes from baseline. SBP will be assessed in accordance with American College of Cardiology/American Heart Association guidelines. Measurements will be taken using an automated oscillometric sphygmomanometer and will be performed in triplicate over the brachial artery of the left arm after 5 minutes of quiet rest, with 1 minute of recovery between measures. SBP will be defined as the average of the 3 pressures.
Change from baseline Nitric Oxide-mediated Endothelial Dependent Dilation (EDD) | EDD will be assessed at baseline and after 6 weeks of training
  Brachial artery Flow Mediated Dilation (BA-FMD), a well-established measure of NO-mediated endothelial function, will be measured by both relative and absolute changes from baseline. BA-FMD will be determined using high-resolution ultrasonography and analyzed with a commercially available software package. An ultrasound probe will be placed 3-6 cm proximal to the antecubital crease on the right arm and a baseline image of the right brachial artery will be obtained. Following baseline, reactive hyperemia will be produced by inflating a rapid-inflating blood pressure cuff. Brachial artery diameter change will be measured for 2 minutes following 5-min of forearm blood flow occlusion.

OTHER OUTCOMES:
Change from baseline proteomic analysis | Proteomics will be performed at baseline and after 6 weeks of training
  Isolated plasma proteins will be subjected to sequential in-solution digestion (Lys-C and trypsin) followed by analysis with tandem mass spectrometry for pre/post changes. Quantitative proteomics using extracted ion abundance, including statistical analysis, will be performed in Progenesis. The resulting quantitative proteomic data sets will be analyzed using DAVID (david.ncifcrf.gov), a well-established tool for gene ontology enrichment analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Dallin Tavoian, PhD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Respiratory and Neurophysiology Laboratory, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available

REFERENCES:
- [Background] Craighead DH, Tavoian D, Freeberg KA, Mazzone JL, Vranish JR, DeLucia CM, Seals DR, Bailey EF. A multi-trial, retrospective analysis of the antihypertensive effects of high-resistance, low-volume inspiratory muscle strength training. J Appl Physiol (1985). 2022 Oct 1;133(4):1001-1010. doi: 10.1152/japplphysiol.00425.2022. Epub 2022 Sep 15. PMID 36107991